CLINICAL TRIAL: NCT05792891
Title: Development of Approaches and Metrics to Measure the Impact and Improve the Clinical Outcomes of Patients With Frailty in the Era of COVID-19.
Brief Title: Approaches and Metrics in Fraily Patients During COVID-19 Era
Acronym: COMETA
Status: Completed | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS1446
Record Dates: First submitted 2023-03-24; First posted 2023-03-31 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-03

CONDITIONS: Frailty; Oncology; Immune Deficiency
MeSH Terms: conditions — Frailty; Neoplasms; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 patients
  Interventions: Other: Collecting biological material from frail patients, with or without COVID-19
- No Covid-19 patients
  Interventions: Other: Collecting biological material from frail patients, with or without COVID-19

INTERVENTIONS:
Other: Collecting biological material from frail patients, with or without COVID-19 — The study planned to collect demographic information, disease history, COVID-19 symptomatology, COVID-19 molecular test details, COVID-19 serological test results, and biobanking of biological specimens (PBMCs, sera, plasma). In addition, clinical analyses, anamnestic data, and pharmacological treatment pieces of information were collected.

SUMMARY:
The COVID-19 pandemic started in December 2019 in Wuhan, the Chinese province of Hubei. Compared to the period of the first epidemic wave (March to May 2020), in the period of the second epidemic wave (October 2020 to July 2021), deceased people have a more significant clinical complexit, as demonstrated by the higher number of comorbidities.The need to allocate significant amounts of healthcare resources to the COVID-19 emergency, deferral of routine healthcare visits, and invitation to avoid medical controls, if not strictly necessary, may have led to interruptions of disease management undersupply of chronic treatments. Consequently, the health status of patients with chronic pathologic conditions have worsened during and beyond the crisis. Patients with cancer, autoimmune disease, and immune deficiencies represented populations with varying immunocompetence, which made translate into higher susceptibility to SARS-CoV-2 and, for this reason, we defined them as frail populations.The main goal of the study was to propel the field of COVID-19 impact on particularly vulnerable categories of patients. The findings of this study could aid in determining the conditions under which healthcare organizations must operate in the event of a pandemic in order to protect patient's rights to care.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for participation in the study
* In the period between April 1, 2021, and September 31, 2022, all COVID-19 positive frail patients identified by molecular swabs taken at participating institutions were included in the study; ii) on a quarterly basis, a cohort of equal numbers of COVID-19 negative frail patients wre identified and paired by disease , gender, and age.

Exclusion Criteria:

* No exclusion criteria were identified

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Frail populations (patients with cancer, autoimmune disease, and immune deficiencies)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Develop general guidelines for clinical care of frail patients | 18 months
  Presence or not of SARS-COV2 infection Presence of specific tumor or HIV-1 infection or psoriasis

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - "Regina Elena" National Cancer Institute, Rome
  - Regina Elena Cancer Institute, Rome

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Silvestris N, Belleudi V, Addis A, Pimpinelli F, Morrone A, Sciacchitano S, Mancini R, Garrisi VM, Costantini M, Ciliberto G, Frisardi V, Piaggio G. Development of Approaches and Metrics to Measure the Impact and Improve the Clinical Outcomes of Patients With Frailty in the Era of COVID-19. The COMETA Italian Protocol. Front Oncol. 2022 Jun 2;12:828660. doi: 10.3389/fonc.2022.828660. eCollection 2022. PMID 35756683